CLINICAL TRIAL: NCT00087022
Title: A Randomized, Double Blind Phase III Study To Evaluate Adjuvant cG250 Treatment Versus Placebo In Patients With Clear Cell RCC And High Risk of Recurrence (ARISER)
Brief Title: Monoclonal Antibody Therapy (Rencarex®) in Treating Patients Who Have Undergone Surgery for Non-metastatic Kidney Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Heidelberg Pharma AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: WX-2003-07-HR; WILEX-WX-2003-07-HR (Other: WILEX); ARISER (Other: WILEX); UCLA-0404015-01 (Other: UCLA); CDR0000372830 (Registry Identifier: PDQ (Physician Data Query)); NCI-2012-00491 (Registry Identifier: CTRP (Clinical Trials Reporting System)); NCT00209183 (obsolete NCT alias)
Record Dates: First submitted 2004-07-08; First posted 2004-07-12 (Estimated); Results first posted 2018-09-12 (Actual); Last update posted 2018-11-27 (Actual); Status verified 2018-10

CONDITIONS: Kidney Cancer
Keywords: clear cell renal cell carcinoma; stage I renal cell cancer; stage II renal cell cancer; stage III renal cell cancer; stage IV renal cell cancer
MeSH Terms: conditions — Kidney Neoplasms; Carcinoma, Renal Cell | interventions — G250 monoclonal antibody

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (Experimental): Patients receive monoclonal chimeric antibody cG250 (synonym names: Rencarex®, girentuximab, and WX-G250) IV over 15 minutes once weekly for 24 weeks.
  Interventions: Biological: girentuximab
- Arm II (Placebo Comparator): Patients receive placebo IV over 15 minutes once weekly for 24 weeks.
  Interventions: Other: placebo

INTERVENTIONS:
Biological: girentuximab — Given IV
  Other Names: Rencarex®, cG250 and WX-G250
  Arms: Arm I
Other: placebo — Given IV
  Arms: Arm II

SUMMARY:
RATIONALE: Monoclonal antibodies can locate tumor cells and either kill them or deliver tumor-killing substances to them without harming normal cells. It is not yet known whether monoclonal antibody therapy is effective in treating kidney cancer.

PURPOSE: This randomized phase III trial is studying monoclonal antibody therapy to see how well it works in treating patients who have undergone surgery for nonmetastatic primary kidney cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Evaluate the disease-free and overall survival of patients with primary clear cell renal cell carcinoma at high risk for recurrence treated with chimeric monoclonal antibody cG250 (WX-G250) vs placebo in an adjuvant setting.

Secondary

* Evaluate the safety of these drugs in these patients.
* Assess the quality of life of patients treated with this drug.
* Perform pharmacokinetic analysis of WX-G250.

OUTLINE: This is a randomized, double-blind, placebo-controlled, multicenter study. Patients are stratified according to risk criteria and participating centers (US vs Non-US). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive monoclonal chimeric antibody cG250 (WX-G250) IV over 15 minutes once weekly for 24 weeks.
* Arm II: Patients receive placebo IV over 15 minutes once weekly for 24 weeks. In both arms, treatment continues in the absence of disease progression or unacceptable toxicity.

Blood samples are collected for pharmacokinetic analysis.

Quality of life is assessed at baseline, at weeks 12 and 24 during treatment, and then at 6 months after completion of study treatment.

Patients are followed every 3 months during years 1 and 2, every 6 months during years 3 and 4, and then annually during year 5 and thereafter.

PROJECTED ACCRUAL: A total of 864 patients out of the expected 856 (428 per treatment arm) were accrued for this trial.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed primary clear cell renal cell carcinoma

  * Meets 1 of the following high risk criteria:

    * T3a, N0/NX, M0 OR T3b, N0/NX, M0 OR T3c, N0/NX, M0 OR T4, N0/NX, M0
    * Any T stage and N + disease and M0
    * T1b, N0/NX, M0 OR T2, N0/NX, M0, each with grade ≥ 3 (Fuhrman or any other nuclear grading system with at least 3 grades)
* Prior nephrectomy (total or partial) of primary renal cell carcinoma with documented clear cell histology within the past 12 weeks

  * No evidence of macroscopic or microscopic residual disease

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-1

Life expectancy

* Not specified

Hematopoietic

* Platelet count > 100,000/mm^3
* WBC > 3,000/mm^3
* Hemoglobin > 10 g/dL

Hepatic

* AST and ALT < 3 times upper limit of normal (ULN)
* Bilirubin < 1.5 times ULN
* Hepatitis B surface antigen (HbsAg) negative
* Hepatitis C antibody negative

Renal

* Creatinine < 2.0 times ULN

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* HIV I and II negative
* No concurrent unrelated illness which can significantly jeopardize patients' clinical status
* No active infection
* No inflammation
* No medical condition or laboratory abnormalities that would preclude study participation
* No other malignancies within the past 5 years except surgically cured nonmelanoma skin cancer or carcinoma in situ of the cervix

PRIOR CONCURRENT THERAPY:

Biologic therapy

* More than 5 years since prior immunotherapy
* No prior murine or chimeric antibody therapy

Chemotherapy

* More than 5 years since prior chemotherapy

Endocrine therapy

* No concurrent corticosteroids above Cushing dose for another disease

  * Physiologic corticosteroid replacement therapy allowed at discretion of the primary investigator

Radiotherapy

* More than 5 years since prior radiotherapy

Surgery

* See Disease Characteristics
* No prior organ transplantation

Other

* No concurrent immunosuppressive agents (e.g., cyclosporine or tacrolimus)

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 864 (Actual)
Dates: Start 2004-07; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pia Kloepfer, MD, Study Director — Heidelberg Pharma AG; Arie Belldegrun, MD, FACS, Principal Investigator — Jonsson Comprehensive Cancer Center
Locations (56):
- United States (39):
  - Anchorage, Alaska
  - Jonsson Comprehensive Cancer Center at UCLA, Los Angeles, California
  - UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - Helen F. Graham Cancer Center at Christiana Hospital, Newark, Delaware
  - Atlantic Urological Associates - Daytona Beach, Daytona Beach, Florida
  - Mayo Clinic - Jacksonville, Jacksonville, Florida
  - Southeastern Research Group, Tallahassee, Florida
  - Winship Cancer Institute of Emory University, Atlanta, Georgia
  - Augusta Oncology Associates - Walton Way, Augusta, Georgia
  - North Idaho Urology - Coeur d'Alene, Coeur d'Alene, Idaho
  - Northeast Indiana Urology, PC, Fort Wayne, Indiana
  - Holden Comprehensive Cancer Center at University of Iowa, Iowa City, Iowa
  - Hematology and Oncology Specialists, LLC - Metairie, Metairie, Louisiana
  - Regional Urology, LLC, Shreveport, Louisiana
  - Feist-Weiller Cancer Center at Louisiana State University Health Sciences, Shreveport, Louisiana
  - Werner-Francis Urology Associates, LLC, Greenbelt, Maryland
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Lahey Clinic Medical Center - Burlington, Burlington, Massachusetts
  - Siteman Cancer Center at Barnes-Jewish Hospital - Saint Louis, St Louis, Missouri
  - Nevada Cancer Institute, Las Vegas, Nevada
  - Community Care Physicians, PC at Urological Institute of NENY, Albany, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - AccuMed Research Associates, Garden City, New York
  - Mount Sinai School of Medicine, New York, New York
  - Hudson Valley Urology, PC, Poughkeepsie, New York
  - Our Lady of Mercy Medical Center Comprehensive Cancer Center, The Bronx, New York
  - Alliance Urology Specialists - Greensboro, Greensboro, North Carolina
  - Carolina BioOncology Institute, Huntersville, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Riverside Methodist Hospital Cancer Care, Columbus, Ohio
  - Urological Associates of Lancaster, Limited, Lancaster, Pennsylvania
  - Urology Associates, Nashville, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - Mary Crowley Medical Research Center at Sammons Cancer Center, Dallas, Texas
  - Urology Associates of South Texas, PA, McAllen, Texas
  - Urology San Antonio, PA - Fredericksburg, San Antonio, Texas
  - Vermont Cancer Center at University of Vermont, Burlington, Vermont
  - CCOP - Virginia Mason Research Center, Seattle, Washington
- Argentina (6):
  - Instituto Alexander Fleming, Cramer, Buenos Aires
  - Hospital Zonal General de Agudos, Ranelagh, Buenos Aires
  - Complejo Medico de la Policia Federal Argentina, Buenos Aires, Buenos Aires F.D.
  - Unidad Oncologica Del Neuquen, Neuquén
  - Centro de Oncologia Rosario, Rosario
  - Clinical Especializada ISIS, Santa Fe
- Brazil (5):
  - Biocancer Centro de Pesq e Trat de Cancer SA, Belo Horizonte, Minas Gerais
  - Nucleo de Oncologia da Bahia, Bahia
  - Instituto Nacional de Cancer, Rio de Janeiro
  - Hospital Sirio-Libanes, São Paulo
  - Universidade Federal de Sao Paulo, São Paulo
- Canada (6):
  - G. Steinhoff Clinical Research, Victoria, British Columbia
  - McMaster Institute of Urology at St. Joseph Healthcare, Hamilton, Ontario
  - Male Health Centre - Oakville, Oakville, Ontario
  - CMX Research, Incorporated, Oakville, Ontario
  - Male Health Centre - North York, Toronto, Ontario
  - Hopital Charles Lemoyne, Greenfield Park, Quebec

REFERENCES:
- [Derived] Chamie K, Donin NM, Klopfer P, Bevan P, Fall B, Wilhelm O, Storkel S, Said J, Gambla M, Hawkins RE, Jankilevich G, Kapoor A, Kopyltsov E, Staehler M, Taari K, Wainstein AJA, Pantuck AJ, Belldegrun AS. Adjuvant Weekly Girentuximab Following Nephrectomy for High-Risk Renal Cell Carcinoma: The ARISER Randomized Clinical Trial. JAMA Oncol. 2017 Jul 1;3(7):913-920. doi: 10.1001/jamaoncol.2016.4419. PMID 27787547
- [Derived] Donin NM, Pantuck A, Klopfer P, Bevan P, Fall B, Said J, Belldegrun AS, Chamie K. Body Mass Index and Survival in a Prospective Randomized Trial of Localized High-Risk Renal Cell Carcinoma. Cancer Epidemiol Biomarkers Prev. 2016 Sep;25(9):1326-32. doi: 10.1158/1055-9965.EPI-16-0226. Epub 2016 Jul 14. PMID 27418270

RESULTS

PARTICIPANT FLOW:
Groups:
- Intervention: Patients receive monoclonal chimeric antibody cG250 (synonym names: Rencarex, girentuximab, and WX-G250) IV over 15 minutes as a single loading dose of 50 mg (week 1) followed by weekly infusions of 20 mg of WX-G250 (weeks 2-24).
  girentuximab: Given IV
- Placebo: Patients receive placebo IV over 15 minutes once weekly for 24 weeks.
  placebo: Given IV
Period: Overall Study
Arm/Group | Intervention | Placebo
Started (ITT Population) | 433 | 431
Treated (Safety Population) | 431 | 424
Completed | 379 | 376
Not Completed | 54 | 55

BASELINE CHARACTERISTICS:
Population: All patients that were enrolled were included in the ITT population used for efficacy analysis; only 855 patients received at least one dose of study treatment and were analyzed for safety (Safety Population, SP)
Groups:
- Intervention: Patients receive monoclonal chimeric antibody cG250 (WX-G250) IV over 15 minutes as a single loading dose of 50 mg (week 1) followed by weekly infusions of 20 mg of WX-G250 (weeks 2-24).
  girentuximab: Given IV
- Total: Total of all reporting groups
Arm/Group | Intervention | Placebo | Total
Number analyzed (Participants) | 433 | 431 | 864
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.2 (9.83) | 57.8 (10.1) | 58.0 (9.98)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 157 | 133 | 290
  Male | 276 | 298 | 574

OUTCOME MEASURES:

1. Primary Outcome: Disease-free Survival
Description: Disease Free Survival (DFS) calculated from the date of randomization up to and including the date of documented relapse as confirmed by the CT, death or start of new anti-tumor therapy.
Time Frame: Until signs of recurrence or until 360 local DFS events have occurred (median follow-up of 4.5 years)
Population: All patients that were enrolled were included in the ITT population used for efficacy analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Placebo
Number analyzed (Participants) | 433 | 431
Participants | 192 | 197
Statistical Analysis 1: Comparison: Intervention vs Placebo; Test type: Superiority; p = 0.737, Log Rank

2. Primary Outcome: Overall Survival
Description: Overall Survival (OS) calculated from the date of randomization to the date of death. Patients with no documented death will be censored at the date of their last study evaluation.
Time Frame: After 419 OS events or 60 months after the last patient has been enrolled, whichever is the later (median follow-up of 4.5 years)
Population: All patients that were enrolled were included in the ITT population used for efficacy analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Placebo
Number analyzed (Participants) | 433 | 431
Participants | 91 | 90
Statistical Analysis 1: Comparison: Intervention vs Placebo; Test type: Superiority; p = 1.012, Log Rank

3. Secondary Outcome: Quality of Life - Global Health Status
Description: Quality of life by EORTC Quality of Life Questionnaire-C30 - Global Health Status at 12 months. A high score for the global health status/QoL represents a high QoL with 0 being the minimum and 100 being the maximum.
Time Frame: At 12 months
Population: Patients still on study who completed the questionnaire
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Placebo
Number analyzed (Participants) | 295 | 315
score on a scale | 71 (21) | 71 (20)

4. Secondary Outcome: Pharmacokinetics of WX-G250
Description: Quantitative determination of cG250 (Girentuximab) trough serum profiles at week 8 (steady state concentration).
Time Frame: Week 8
Population: Patients who did sign amendment #3 to the study protocol and received their cG250 infusion as scheduled in the study protocol
Measure: Mean (Standard Deviation); unit: µg/mL
Arm/Group | Intervention
Number analyzed (Participants) | 340
µg/mL | 8.7 (5.8)

5. Post Hoc Outcome: Disease Free Survival (DFS) for Patients With CAIX Score >= 2.6
Description: This analysis includes patients having a CAIX Expression equal or above the CAIX score of 2.6.
  The CAIX score is determined on the basis of CAIX expression via immunohistochemistry described by a combination of tumor cell extent and staining intensity.
  Disease Free Survival (DFS) calculated from the date of randomization up to and including the date of documented relapse as confirmed by the CT, death or start of new anti-tumor therapy.
Time Frame: Until signs of recurrence or until 360 local DFS events have occurred (median follow-up of 4.5 years)
Population: This analysis includes patients having a CAIX Expression equal or above the CAIX score of 2.6.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Placebo
Number analyzed (Participants) | 69 | 82
Participants | 20 | 39
Statistical Analysis 1: Comparison: Intervention vs Placebo; Test type: Superiority; p = 0.022, Log Rank

ADVERSE EVENTS:
Arm/Group | Intervention | Placebo
Serious Adverse Events (participants affected / at risk) | 36/431 | 36/424
Other Adverse Events (participants affected / at risk) | 164/431 | 166/424
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Intervention (N=431) | Placebo (N=424)
ANAEMIA (Blood and lymphatic system disorders) | 1 | 0
LYMPHADENOPATHY (Blood and lymphatic system disorders) | 1 | 0
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 1 | 1
ATRIAL FIBRILLATION (Cardiac disorders) | 1 | 0
CARDIAC FAILURE (Cardiac disorders) | 0 | 1
CHEST DISCOMFORT (Cardiac disorders) | 0 | 1
MYOCARDIAL INFARCTION (Cardiac disorders) | 2 | 1
ABDOMINAL ADHESIONS (Gastrointestinal disorders) | 1 | 0
ASCITES (Gastrointestinal disorders) | 1 | 0
DIARRHOEA (Gastrointestinal disorders) | 0 | 1
DUODENAL ULCER PERFORATION (Gastrointestinal disorders) | 0 | 1
GASTRIC ULCER (Gastrointestinal disorders) | 1 | 1
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 1 | 0
OESOPHAGITIS (Gastrointestinal disorders) | 1 | 0
PANCREATITIS ACUTE (Gastrointestinal disorders) | 1 | 0
CHEST PAIN (General disorders) | 0 | 1
BILIARY DILATATION (Hepatobiliary disorders) | 1 | 0
CHOLECYSTITIS CHRONIC (Hepatobiliary disorders) | 0 | 1
BRONCHITIS (Infections and infestations) | 0 | 1
CYSTITIS (Infections and infestations) | 0 | 1
EMPYEMA (Infections and infestations) | 0 | 1
ERYSIPELAS (Infections and infestations) | 0 | 1
ESCHERICHIA SEPSIS (Infections and infestations) | 1 | 0
PNEUMONIA (Infections and infestations) | 0 | 2
POSTOPERATIVE ABSCESS (Infections and infestations) | 0 | 1
PYELONEPHRITIS (Infections and infestations) | 1 | 0
SINUSITIS (Infections and infestations) | 1 | 0
FEMUR FRACTURE (Injury, poisoning and procedural complications) | 1 | 0
INCISIONAL HERNIA (Injury, poisoning and procedural complications) | 0 | 1
MENISCUS LESION (Injury, poisoning and procedural complications) | 1 | 0
PELVIC FRACTURE (Injury, poisoning and procedural complications) | 1 | 0
POST PROCEDURAL HAEMORRHAGE (Injury, poisoning and procedural complications) | 1 | 0
THERMAL BURN (Injury, poisoning and procedural complications) | 0 | 1
BIOPSY LUNG (Investigations) | 0 | 1
MEDIASTINOSCOPY (Investigations) | 0 | 1
DEHYDRATION (Metabolism and nutrition disorders) | 0 | 1
DIABETES MELLITUS (Metabolism and nutrition disorders) | 0 | 1
HYPOGLYCAEMIA (Metabolism and nutrition disorders) | 0 | 1
BACK PAIN (Musculoskeletal and connective tissue disorders) | 1 | 1
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 0 | 1
PATHOLOGICAL FRACTURE (Musculoskeletal and connective tissue disorders) | 0 | 1
BREAST CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
LUNG NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
METASTASES TO CENTRAL NERVOUS SYSTEM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
METASTASES TO LUNG (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
METASTASES TO LYMPH NODES (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
OVARIAN CYST (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
PROSTATE CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2
RECURRENT CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
SALIVARY GLAND CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
THYROID NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
CEREBRAL HAEMORRHAGE (Nervous system disorders) | 1 | 0
HEADACHE (Nervous system disorders) | 1 | 1
PERIPHERAL NERVE LESION (Nervous system disorders) | 0 | 1
PREGNANCY (Pregnancy, puerperium and perinatal conditions) | 0 | 1
HAEMATURIA (Renal and urinary disorders) | 1 | 1
RENAL FAILURE ACUTE (Renal and urinary disorders) | 1 | 0
URINARY RETENTION (Renal and urinary disorders) | 0 | 1
OVARIAN MASS (Reproductive system and breast disorders) | 1 | 0
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 0 | 1
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 2 | 2
PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 1 | 0
COLON POLYPECTOMY (Surgical and medical procedures) | 0 | 1
MALIGNANT TUMOUR EXCISION (Surgical and medical procedures) | 1 | 0
RENAL TUMOUR EXCISION (Surgical and medical procedures) | 1 | 0
THYROID OPERATION (Surgical and medical procedures) | 0 | 1
DEEP VEIN THROMBOSIS (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Intervention (N=431) | Placebo (N=424)
DIARRHOEA (Gastrointestinal disorders) | 27 | 39
NAUSEA (Gastrointestinal disorders) | 35 | 29
VOMITING (Gastrointestinal disorders) | 28 | 18
BACK PAIN (Musculoskeletal and connective tissue disorders) | 34 | 37
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 27 | 22
NASOPHARYNGITIS (Infections and infestations) | 30 | 33
FATIGUE (General disorders) | 28 | 39
ASTHENIA (General disorders) | 19 | 22
HEADACHE (Nervous system disorders) | 40 | 39
HYPERTENSION (Vascular disorders) | 34 | 25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less